CLINICAL TRIAL: NCT00732706
Title: Femoral Nerve Block: Anatomical Insertion Point - A Prospective Randomised Double-Blind Controlled Trial
Acronym: FNB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. Imad Awad, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SHSCHOACFNB
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Femoral Nerve Disease
Keywords: FNB; Femoral Nerve; Sartorius Twitch; Quadriceps Twitch; Analgesia; Anesthesia
MeSH Terms: conditions — Femoral Neuropathy; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sartorius Twitch (Other): Femoral Nerve detection using Sartorius Twitch
  Interventions: Procedure: Sartorius Muscle Twitch
- Quadriceps Twitch (Other): Femoral Nerve detection using Quadriceps Twitch
  Interventions: Procedure: Quadriceps Muscle Twitch

INTERVENTIONS:
Procedure: Sartorius Muscle Twitch — Stimulation of the femoral nerve branch responsible for activating the Sartorius Muscle fascia with the lowest possible current.
  Arms: Sartorius Twitch
Procedure: Quadriceps Muscle Twitch — Stimulation of the femoral nerve branch responsible for activating the Quadriceps Muscle fascia with the lowest possible current.
  Arms: Quadriceps Twitch

SUMMARY:
Nerve blocks are an effective way to control pain after surgery. There are two major nerves that provide sensation to the knee: the femoral nerve provides sensation to the front of the knee and sciatic nerve provides sensation to the back of the knee. The femoral nerve has two branches. To locate the nerve, we use a machine called (Nerve stimulator) which is attached to the needle used for nerve block. Use of a nerve stimulator is standard practice for this procedure. Ultrasound is being increasingly used to locate nerves but is not used universally. We will use the nerve stimulator and ultrasound to locate the femoral nerve but patients will randomly be selected to enter a group looking at the stimulation of one or the other branches of the femoral nerve. The two branches when stimulated produce different muscle contractions in the thigh. We do not know from research which is the optimal contraction to position the needle to get the best block. After the knee replacement patients will still have the same analgesic medication available as patients would have received if they were not in the study.

DETAILED DESCRIPTION:
To determine if needle insertion at the inguinal crease with stimulation of sartorius muscle (anterior branch) causes an equivalent block to the classical method with stimulation of the quadriceps femoris muscle (posterior branch), for femoral nerve blockade. To test this hypothesis, we plan to conduct a randomised controlled double-blind study comparing success of femoral never block (motor and sensory) using sartorius twitch versus quadriceps femoris twitch as an end point.

We will also evaluate the local anesthetic distribution under the facia iliaca sheath using ultrasound imaging.

Methods: Following institutional ethical approval and obtaining written informed consent, we plan to recruit 60 patients aged 18-80, ASA I-III scheduled to undergo unilateral total knee arthroplastly in this prospective, randomised, double blinded controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80
* ASA Status I-III
* Unilateral total knee arthroplasty Patients

Exclusion Criteria:

* Patients with a history of significant medical or psychiatric problems
* Patients with BMI > 35
* Unable to cooperate with the study protocol or unable to understand English
* Had allergy to local anaesthetics or fentanyl
* Prior surgery in the inguinal region
* Sensory or motor disease
* Diabetic neuropathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Comparing success of femoral never block (motor and sensory) using sartorius twitch versus quadriceps femoris twitch as an end point, using Motor and Sensory Scores. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Imad Awad, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada